CLINICAL TRIAL: NCT05261945
Title: The Effects of Manual Therapy Versus Stretching Exercise Versus Routine Physical Therapy on Work-related Pain, Among Patients With Non-specific Chronic Neck Pain Working as Chefs: A Randomised Controlled Trial
Brief Title: Effects of Manual Therapy Versus Stretching Exercise Versus Routine Physical Therapy on Work-related Pain, Among Chefs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-FSD-00297
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Neck Pain
Keywords: Manual Therapy; Stretching Exercises; Routine Physical Therapy; Non Specific Chronic Neck Pain; Restaurant Chefs
MeSH Terms: conditions — Neck Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Our study will be double-blinded, outcome assessor-blinded and patient- blinded. The assessor will be blinded to avoid being biased during the outcome assessment. And, participants will be blinded to avoid the their incompliance during sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Routine Physical Therapy (Experimental): 1. Electrotherapy
  2. Exercises.
     * Electrotherapy Hot pack Patients will be in prone position and for relaxation pillow will place beneath the abdomen. Then to reduce muscle spasm and to induce vasodilation hot pack will use for 15 minutes. Treatment with hot pack helps in improving and relaxing the muscle spasm and soft tissue elasticity.
  TENS TENS will be of 50 Hz, duration of pulse will be<150 microseconds, for 15 minutes to reduce pain.
  TENS and Hot Pack will use at the same time for 15 minutes.
  Ultrasound Ultrasound's gel will be applied on outer surface of skin with 2-3 mm thickness. Then ultrasound which frequency will be 1MHz applied for 5 min.
  • Exercises Passive Range of Motion exercises for 10 minutes
  1. Neck Flexion
  2. Neck Side bending
  3. Neck Rotation
  4. Isometric neck flexion
  5. Isometric neck extension
  6. Isometric neck side bending
  These exercises will repeat 3 times within the treatment program.
  Interventions: Other: Routine Physical Therapy
- Manual Therapy And Routine Physical Therapy (Experimental): The routine physical therapy will be applied first, in which electrotherapy will applied for 20 mins, TENS and hot pack for 15 mins, ultrasound for 5 mins.
  Manual therapy
  Natural Apophyseal Glides The natural apophyseal glides, which will be applied between C2 and C7, will be the Manual Muscle Testings first action. Patients may request to sit and lean on a chair. The oscillatory motions will reapply the mobilization.
  Sustained Natural Apophyseal Glides Sustained Natural Apophyseal Glides will be a mixture of mobilization and active gestures/movements.
  5 repetitions for 10 minutes of each.
  Interventions: Other: Manual Therapy And Routine Physical Therapy
- Stretching Exercises And Routine Physical Therapy (Experimental): The routine physical therapy will be applied first, in which electrotherapy will applied for 20 minutes, TENS and hot pack is applied for 15 minutes at the same time, then ultrasound will applied for 5 minutes.
  Stretching exercises will be done in the following order;
  For trapezius: Stretching into lateral flexion for the upper part, For scalene: rotation and ipsilateral flexion For the extensor muscles: flexion will be performed.
  Performing each action for 30 seconds with 5 repetitions for 10 minutes Finally, by retruding the jaw, a neck straightening exercise can be performed.
  Interventions: Other: Stretching Exercises And Routine Physical Therapy

INTERVENTIONS:
Other: Routine Physical Therapy — Routine Physical Therapy treatment with hot pack, TENS, and ultrasound helps in improving and relaxing the muscle spasm and soft tissue elasticity along pain reduction.
  Arms: Routine Physical Therapy
Other: Manual Therapy And Routine Physical Therapy — Mulligan is consider one of the most effective technique of mobilization.it is also important treatment for neck pain so that many physiotherapist used mulligan by including several methods such as Natural Apophyseal Glides or Sustained Natural Apophyseal Glides.
  Arms: Manual Therapy And Routine Physical Therapy
Other: Stretching Exercises And Routine Physical Therapy — Regular stretching helps increase your range of motion in the joints, improves blood circulation and posture and alleviates muscular tension throughout the body.
  Arms: Stretching Exercises And Routine Physical Therapy

SUMMARY:
The aim of this research is to analyze the effect of Mulligan technique versus stretching techniques and versus routine physical therapy on pain, range of motion and functional disability among restaurant chefs presenting with non-specific chronic pain.

DETAILED DESCRIPTION:
A Randomized Control Trail study will be conducted, at Riphah International University Faisalabad after the approval of synopsis. Purposive sampling will be used to enroll the patients. Patients will be selected according to the pre-defined inclusion and exclusion criteria. The patients who will meet the inclusion criteria are allocated into three groups. The patients of group A will receive Routine physical therapy only. Group B will receive manual therapy and routine physical therapy while Group C will receive stretching exercises and routine physical therapy. The outcomes will be measured by the Neck Disability Index, visual analogue scale and bubble inclinometer. The data of patients will be recorded pre-treatment and post-treatment. The comparison between pre-treatment and post-treatment data will be done after 3 months. Informed consent will be taken from each patient. Data entry and analysis will be done with Statistical Package of Social Sciences Version 20 software.

ELIGIBILITY:
Inclusion Criteria:

* For at least 3 months, you've been suffering from neck pain
* Any Neurological problems
* For the previous three months, the patient has taken some analgesic drug for neck pain.
* Rheumatological issues
* Non-specific neck pain
* Age 18-60 years

Exclusion Criteria:

Neck pain due to,

* Tumors
* Ankylosing Spondylitis
* Fracture
* Dislocation
* Cord compression
* Insufficiency of the vertebrobasilar artery
* Osteoprosis
* Anticoagulant or corticosteroid therapy for a long period of time
* Pain due to any congenital deformity, inflammation or any infection
* Carcinoma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | 12th Week
  A Visual Analogue Scale is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.
Neck disability index | 12th Week
  The Neck Disability Index is a 10-item questionnaire that measures a patient's self-reported neck pain related disability. A higher Neck Disability Index score means the greater a patient's perceived disability due to neck pain
Bubble inclinometer | 12th Week
  The Bubble Inclinometer precisely measures, tests and evaluates the ranges of motion of neck. While using, place the Inclinometer near the joint to be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No